CLINICAL TRIAL: NCT04036279
Title: A Prospective, Multicenter, Clinical Outcome Study of the NANOS Neck Preserving Stem in Patients With Degenerative Hip Joint Disease
Brief Title: NANOS Neck Preserving Hip Stem
Acronym: NANOS
Status: Terminated | Type: Observational
Why Stopped: This study was originally designed to meet MDR commitments. MDR Approval was secured without this study. Therefore, this study does not fulfil its role as a regulatory body commitment.
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Other Study IDs: R11014-1
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Primary Osteoarthritis; Secondary Osteoarthritis; Dysplasia Osteoarthritis; Avascular Femoral Neck Necrosis; Post-Traumatic Femoral Neck Necrosis; Intact Femoral Neck With Good Bone Quality
Keywords: NANOS; Hip; Neck Preserving Stem
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Total Hip Arthroplasty

SUMMARY:
The objective of this study is to determine the long-term safety and effectiveness of the NANOS neck preserving stem in terms of radiographic and clinical performance as well as short-, mid- and long-term survivorship

DETAILED DESCRIPTION:
The goal of this multicenter clinical observation is to validate short-, mid-, and long-term outcome (efficacy and safety) of the NANOS neck preserving hip stem.

Effectiveness Measures:

* Evaluation of function, range of motion (ROM) and pain as assessed by Harris Hip Score, HOOS Score [4-6], UCLA Activity Rating [7]
* Radiographic changes as defined by radiolucent lines, osteolysis, hypo- and hypertrophy, implant loosening or migration

Safety evaluations:

* Intra- and peri-operative device-related adverse events (AE) and complications up to discharge
* Postoperative AE up to 10 years

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:
* Patient requires Primary total hip replacement (THR) to the affected side, unilateral or bilateral. Bilateral only if >3 months after the first THR
* Patient agreed to participate in the MCO study by signing the Informed Consent form.
* Age of patient at date of surgery 18 to 65 years
* Patient is likely to comply with study follow-up requirements

Exclusion criteria:

* Previously failed endoprosthesis and /or THR components in relevant hip
* Patient has proven osteoporosis
* Pronounced coxa valga with a femoral neck angle > 145º
* Pronounced coxa vara with a femoral neck angle < 125º
* History of infection in the affected joint; systemic infections
* Grossly insufficient femoral or acetabular bone stock in the involved hip where a revision cup is indicated
* Spinal disease with neurologic movement disorders
* Alcoholism or addictive disorders
* ASA score is 3 or 4
* Body mass index (BMI) > 30
* Patient is pregnant or being pregnant during follow up intervals
* Patients understanding of the language is insufficient for understanding the Patient Information and Consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinic for Orthopedics
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2010-01-21 (Actual); Primary Completion 2023-03 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
Long term survivorship of Nanos | 10 years
  Revision for any reason. Implant survivorship at 10 years post study procedure. A revision is a surgical procedure of the study hip where one or more of the study components are removed and replaced with new implants

OTHER OUTCOMES:
Intra- and peri-operative device-related adverse events (AE) and complications up to discharge | 10 years
  Any reported safety events or complications up to 10 years post study procedure
Postoperative AE up to 10 years | 10 years
  Any reported safety events or complications up to 10 years post study procedure
Evaluation of function, range of motion and pain assessed by Harris Hip Score | 10 years
  Harris Hip Score is a joint specific score that consists of 10 items covering domains of pain (1 item, 0-44 points), function (7 items, 0-47 points), functional activities, absence of deformity (1 item, 0 or 4 points), and hip range of motion (2 items, 0-5 points). Scores range from 0 (worst) to 100 (best).
  HHS scores for each subject will further be categorized as follows: Excellent (90-100); Good (80-89); Fair (70-79); Poor (60-69) and; Very poor (<60).
Evaluation of function, range of motion and pain as assessed by HOOS score | 10 years
  HOOS consists of 5 subscales: Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and hip related QOL. The last week is taken into consideration when answering the questions. Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Evaluation of function, range of motion and pain as assessed by UCLA Activity Rating | 10 years
  UCLA Activity Score is a measure of physical activity levels in subjects undergoing total joint arthroplasty. The scale is from 1 - 10 with higher values indicating greater physical function.
Radiographic changes as defined by resorption, radiolucent lines, osteolysis, hypo- and hypertrophy, implant migration or loosening | 10 years
  Any radiographic changes up to 10 years post study procedure

CONTACTS AND LOCATIONS:
Overall Officials: Turgay Efe, Dr.med, Principal Investigator — Phillips University Marburg, Germany
Locations (3):
- University Marburg, Orthopedics and Rheumatology, Marburg, Germany
- Medisch Centrum Alkmaar, Alkmaar, Netherlands
- Samodzielny Publiczny Wojewodzki Spital, Piekary Śląskie, Poland

IPD SHARING:
Plan to Share IPD: No